CLINICAL TRIAL: NCT01841515
Title: Effect of Desmopressin on Platelet Function in CKD Patients on Antiplatelet Agent Who Need Emergent Temporary Catheter Insertion for Hemodialysis
Brief Title: Effect of Desmopressin on Platelet Function in CKD Patients on Antiplatelet Drug
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Ulsan (Other)
Responsible Party: Principal Investigator, Soon Bae Kim, M.D., PhD., Professor of Medicine, University of Ulsan
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCT00134031
Record Dates: First submitted 2013-04-23; First posted 2013-04-26 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Bleeding; Tachycardia; Dyspnea
MeSH Terms: conditions — Hemorrhage; Tachycardia; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Desmopressin (Experimental): Twenty five patients with chronic kidney disease and who were taking antiplatelet agents and needed an emergent catheter insertion for hemodialysis
  Interventions: Drug: Desmopressin administration

INTERVENTIONS:
Drug: Desmopressin administration

SUMMARY:
Prolonged Collagen/Epinephrine - closure time (CEPI-CT) indicates platelet dysfunction in CKD patients taking antiplatelet agent. The synthetic vasopressin derivative, Desmopressin (DDAVP) shortens the prolonged bleeding time and improves platelet dysfunction measured by in vitro closure time: CEPI-CT in uremic patients. Desmopressin also antagonizes the in vitro platelet dysfunction induced by GPIIb/IIIa inhibitors, clopidogrel and aspirin. The investigators designed a prospective study to evaluate the effect of desmopressin on platelet function, as measured by in vitro collagen/epinephrine - closure time, in uremic patients who were taking antiplatelet drugs.

ELIGIBILITY:
Inclusion Criteria:

* adult uremic patients with one or more antiplatelet medication,
* prolonged collagen/epinephrine (CEPI) closure time,
* need for emergent hemodialysis and
* subsequent catheter insertion

Exclusion Criteria:

* acute coronary syndrome,
* hemophilia, and nephrogenic diabetes insipidus,
* allergy against desmopressin

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
collagen-epinephrine closure time | 1 hour
  In vitro closure time (CT), measured using a platelet function analyzer (PFA)-100, is a relatively new tool for investigation of primary hemostasis. This system has been shown to be efficacious in evaluating abnormalities of primary hemostasis.

SECONDARY OUTCOMES:
Bleeding after procedure | 1-4 hr after procedure
  we observe incidence of bleeding complication after procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea